CLINICAL TRIAL: NCT04092127
Title: Pain Quantification Study During a Screening for Retinopathy of Premature Babies by RetCam
Brief Title: Pain of Premature Babies and RetCam (DOLICAM)
Acronym: DOLICAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.172; 2019-A01982-55 (Other: ID RCB)
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Premature Infant Disease; Retinopathy of Prematurity
Keywords: RetCam; Pain evaluation; PIPP (Premature Infant Pain Profile) Score; Screening for Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature infants (<32 weeks of Gestation Age): premature babies (<32 weeks of Gestation Age) to be screened with RetCam for retinopathy of prematurity and who will be filmed during the screening procedure to evaluate pain with the PIPP score (Premature Infant Pain Profile)
  Interventions: Other: Video Record

INTERVENTIONS:
Other: Video Record — Video Record of the premature infant face before and during the RetCam screening of retinopathy of prematurity

SUMMARY:
It is a single-center prospective observational descriptive study.

studied population is premature infants, hospitalized in the neonatology department of the University Hospital of Grenoble and for whom the RetCam examination is planned for screening for retinopathy of prematurity if they are at risk (prematurity <32 weeks).

To measure their pain during the examination, it will be a matter of filming the face of the child for 15 seconds before the examination, then 2 times 30 seconds at two distinct times. The PIPP (Premature Infant Pain Profile) score includes a percentage of time on these 30 seconds where 3 items are found modified and a monitoring of heart rate and oxygen saturation.This time calculation can not be done live and requires video recording of the child's face during the exam.

The statistical analyzes will be adjusted for sex, gestational age at birth, weight, and pain from birth (determined by the number of doses of level 1 analgesics received by the baby and the number of days (from birth to to the RetCam examination) when the baby received > level 1 analgesics).

DETAILED DESCRIPTION:
It is a single-center prospective observational descriptive study.

The studied children will be premature infants hospitalized in the neonatology department of the University Hospital of Grenoble and for whom the RetCam examination is planned for screening for retinopathy of prematurity if they are at risk (prematurity <32 weeks). These exams fit into a routine care.

To measure their pain during the examination, it will be a matter of filming the face of the child for 15 seconds before the examination, then 2 times 30 seconds at two distinct times.

The PIPP (Premature Infant Pain Profile) score includes a percentage of time on these 30 seconds where 3 items are found modified and a monitoring of heart rate and oxygen saturation. (Please note that the recording of the constants of the child is already integrated into the current care in the neonatology department of the University Hospital of Grenoble and will not be added for the purpose of the study.) Expected scores should be about 12/21, despite the use of analgesic agent.

This time calculation can not be done live and requires video recording of the child's face during the exam. After parental information and non-opposition consent of the parents, the child can be filmed and his constants annotated during the current care. Parents can attend this observational procedure.

The statistical analyzes will be adjusted for sex, gestational age at birth, weight, and pain from birth (determined by the number of doses of level 1 analgesics received by the baby and the number of days (from birth to to the RetCam examination) when the baby received > level 1 analgesics).

ELIGIBILITY:
Inclusion Criteria:

* Premature born before 31 weeks of Gestational Age or birth weight less than 1250 grams or less than 1300 grams and less than 33 weeks of Gestational age, with risk factor (prolonged oxygen therapy, sepsis, prolonged use of inotropes)
* Corrected age above 31 weeks of gestational age at the time of inclusion
* Having to do a RetCam exam in the neonatology department of the University Hospital of Grenoble.
* No opposition of the subject's parents

Exclusion Criteria:

* Subject under guardianship or subject deprived of liberty
* Premature requiring a respiratory aid limiting the observation of the face at the time of the examination.
* Non-compliance with the analgesic protocol of the service, prior to examination (paracetamol and sugar solutions).
* Prematurity with a facial malformation and / or neurological disorder that prevents the rating of pain by the PIPP scale

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The studied population corresponds to the premature infants of more than 31 weeks of gestational age and of more than 4 weeks of life, which require a retinopathy of the premature screening by RetCam in the service of neonatology, neonatal resuscitation of the University Hospital of Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Pain quantification with the PIPP (Premature Infant Pain Profile) scale during a screening for retinopathy of prematurity with RetCam (with the analgesic protocol set up in the neonatology department of the University Hospital of Grenoble) | during the screening of retinopathy of prematurity by RetCam
  the highest value of pain assessment by the PIPP (Premature Infant Pain Profile) scale during the RetCam exam. The 2 assessments will be done:
  * after eyelid speculum placement (30 seconds evaluation)
  * after RetCam installation (30s)
  PIPP: the higher is the score, the higher the pain is.
  Total score (from 0 to 21) = addition of 7 subscores (0-3):
  * Gestational Age: 36 weeks or more / 32-35 weeks + 6 days / 28-31 weeks + 6 days / Less than 28 weeks
  * Behavioural State: Active, awake, eyes open, facial, movement / Quiet awake, eyes open, no facial movements / Active sleep, eyes closed, facial movements / Quiet sleep, eyes closed, no facial movements
  * heart rate maximum: 0 bpm (beats per minute) increase / 5-15 bpm increase / 15-24 bpm increase / 25+ bpm increase.
  * oxygen saturation minimum: 92-100%/89-91%/88-85%/<85%
  * Brow Bulge: None/Minimum/Moderate/Maximum
  * Eye Squeeze: None/Minimum/Moderate/Maximum
  * Naso-labial furrow: None/Minimum/Moderate/Maximum

SECONDARY OUTCOMES:
Determination of the most painful part of the examination : Comparison of the pain felt when the eyelid speculums are placed and the pain felt during during the examination by the RetCam (during the same gesture). | during the usual care procedure of screening of retinopathy of prematurity by RetCam
  Numerical value of PIPP 30 seconds after eyelid speculum placement compared to the PIPP numerical value of 30 seconds after the start of the camera examination.
  PIPP: the higher is the score, the higher the pain is.
  Total score (from 0 to 21) = addition of 7 subscores (0-3):
  * Gestational Age: 36 weeks or more / 32-35 weeks + 6 days / 28-31 weeks + 6 days / Less than 28 weeks
  * Behavioural State: Active, awake, eyes open, facial, movement / Quiet awake, eyes open, no facial movements / Active sleep, eyes closed, facial movements / Quiet sleep, eyes closed, no facial movements
  * heart rate maximum: 0 bpm (beats per minute) increase / 5-15 bpm increase / 15-24 bpm increase / 25+ bpm increase.
  * oxygen saturation minimum: 92-100%/89-91%/88-85%/<85%
  * Brow Bulge: None/Minimum/Moderate/Maximum
  * Eye Squeeze: None/Minimum/Moderate/Maximum
  * Naso-labial furrow: None/Minimum/Moderate/Maximum

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Debillon, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jefferies AL; Canadian Paediatric Society, Fetus and Newborn Committee. Retinopathy of prematurity: An update on screening and management. Paediatr Child Health. 2016 Mar;21(2):101-8. doi: 10.1093/pch/21.2.101. PMID 27095887
- [Result] Chiang MF, Melia M, Buffenn AN, Lambert SR, Recchia FM, Simpson JL, Yang MB. Detection of clinically significant retinopathy of prematurity using wide-angle digital retinal photography: a report by the American Academy of Ophthalmology. Ophthalmology. 2012 Jun;119(6):1272-80. doi: 10.1016/j.ophtha.2012.01.002. Epub 2012 Apr 27. PMID 22541632
- [Result] Ezz El Din ZM, El Sada MA, Ali AA, Al Husseiny K, Yousef AA. Comparison of digital imaging screening and indirect ophthalmoscopy for retinopathy of prematurity. Indian J Pediatr. 2015 Jan;82(1):80-3. doi: 10.1007/s12098-014-1525-1. Epub 2014 Aug 1. PMID 25081804
- [Result] Disher T, Cameron C, Mitra S, Cathcart K, Campbell-Yeo M. Pain-Relieving Interventions for Retinopathy of Prematurity: A Meta-analysis. Pediatrics. 2018 Jul;142(1):e20180401. doi: 10.1542/peds.2018-0401. Epub 2018 Jun 1. PMID 29858451
- [Result] Ranger M, Grunau RE. Early repetitive pain in preterm infants in relation to the developing brain. Pain Manag. 2014 Jan;4(1):57-67. doi: 10.2217/pmt.13.61. PMID 24641344
- [Result] Vinall J, Grunau RE. Impact of repeated procedural pain-related stress in infants born very preterm. Pediatr Res. 2014 May;75(5):584-7. doi: 10.1038/pr.2014.16. Epub 2014 Feb 5. PMID 24500615
- [Result] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Result] Stevens B, Johnston C, Taddio A, Gibbins S, Yamada J. The premature infant pain profile: evaluation 13 years after development. Clin J Pain. 2010 Nov-Dec;26(9):813-30. doi: 10.1097/AJP.0b013e3181ed1070. PMID 20717010